CLINICAL TRIAL: NCT00518453
Title: A Phase II, Open-Label, Uncontrolled, Single Center Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated Influenza Vaccine Ph.Eur, Formulation 2007-2008, When Administered to Non-Elderly Adult and Elderly Subjects
Brief Title: Immunogenicity of a Surface Antigen, Inactivated Influenza Vaccine Formulation 2007-2008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V78P5S; 2007-002063-27
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: Fluvirin (Experimental)
  Interventions: Biological: Surface antigen inactivated influenza vaccine

INTERVENTIONS:
Biological: Surface antigen inactivated influenza vaccine — 1 dose of Fluvirin 2007/2008 Northern Hemisphere vaccine composition

SUMMARY:
Due to antigenic changes of influenza viruses, the virus strains used in influenza vaccines are adjusted every year according to WHO and CPMP recommendations. Immunogenicity and tolerability of the newly composed vaccines are subject for evaluation in a yearly clinical trial in non-elderly adults and elderly subjects (CPMP/BWP/214/96).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects eligible for enrollment into this study are male and female adult volunteers

Exclusion Criteria:

* Any serious disease

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
evaluate the antibody response to each influenza vaccine antigen | 21 days post-immunization

SECONDARY OUTCOMES:
Safety and tolerability of the study vaccine in the study population | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- The Health Centre, Suffolk, United Kingdom